CLINICAL TRIAL: NCT00596388
Title: Usage of the Home Macular Perimeter (HMP) in Intermediate Age Related Macular Degeneration Patients Pilot Study
Brief Title: Usage of the Home Macular Perimeter (HMP)
Acronym: HMP
Status: Completed | Type: Observational
Sponsor: Notal Vision Ltd. (Industry)
Responsible Party: Sponsor
Organization: Notal Vision Inc. (Industry)
Other Study IDs: HMP-PU1; 0197-07
Record Dates: First submitted 2008-01-07; First posted 2008-01-17 (Estimated); Last update posted 2013-05-15 (Estimated); Status verified 2013-05

CONDITIONS: Age Related Macular Degeneration
Keywords: HMP, AMD, CNV, PHP, HPHP
MeSH Terms: conditions — Macular Degeneration; Choroidal Neovascularization

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Subjects diagnosed as intermediate AMD

SUMMARY:
Demonstrate the ability of the current interactive tutorial and 1-800 support to teach an AMD patient to use the HMP device.

DETAILED DESCRIPTION:
The pilot study purpose is to demonstrate that the tutorial which is part of the device software, is giving sufficient training for the intended users.

ELIGIBILITY:
Inclusion Criteria:

* Capable and willing to sign a consent form and participate in the study
* Subjects diagnosed as intermediate AMD in at least one eye
* Age >50 years
* VA with habitual correction >20/60 in the study eye
* Ability to speak, read and understand instructions in Hebrew
* Familiar with computer usage

Exclusion Criteria:

* Evidence of macular disease other than AMD or glaucoma in the study eye
* Presence of any significant media opacity that precludes a clear view of the macular area as identified in the study eye by biomicroscopy, CFP.
* Any non-macular related ocular surgery performed within 3 months prior to study entry in the target eye
* Participation in another study with the exclusion of AREDS study
* Patients diagnosed with geographic atrophy (GA)

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: • Subjects diagnosed as intermediate AMD
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2008-03; Primary Completion 2013-01 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects who manage to use the device as in a daily testing | 6 month

CONTACTS AND LOCATIONS:
Overall Officials: Yaron Mr Lang, MD, Principal Investigator — Haemek Hospital
Locations (1):
- Haemek Medical center, Afula, Israel

REFERENCES:
- See also: sponsor site — http://www.notalvision.com